CLINICAL TRIAL: NCT01239771
Title: A Phase I, Double-blind, Placebo-controlled, Parallel Group Study to Assess the Safety, Tolerability and Pharmacokinetics of TC-5214 Given as Multiple Ascending Oral Doses in Medically Stable Elderly Subjects
Brief Title: A Study to Assess Safety and Tolerability as Well as Absorption and Excretion of TC-5214 in Medically Stable Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D4130C00013
Record Dates: First submitted 2010-10-28; First posted 2010-11-11 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2011-01

CONDITIONS: Elderly Subjects 65 Years and Older, Healthy or With a Stable Disease and Treatment.
Keywords: Safety; tolerability; healthy; stable disease; oral; tablet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): TC-5214
  Interventions: Drug: TC-5214
- 2 (Placebo Comparator): Placebo matched to TC-5214
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TC-5214 — Tablet 1, 2, or 4 mg of TC-5213 will be given twice daily for 4 days and once on the 5th day.
  Arms: 1
Drug: Placebo — Two subjects in each cohort will be given placebo.
  Arms: 2

SUMMARY:
The purpose of the study is to assess safety, tolerability and pharmacokinetics of TC-5214 in medically stable elderly subjects following multiple oral doses.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable male and female subjects aged greater than or equal to 65 years with suitable veins for cannulation or repeated venipuncture. Subjects may have controlled chronic diseases such as hypertension, type 2 diabetes, osteoarthritis, stable chronic obstructive pulmonary disease, mild or moderate renal insufficiency (Estimated glomerular filtration rate (eGFR) per the Modified Diet in Renal Disease [MDRD] formula >50 mL/min/1.73 m2), rhinitis etc. as long as there has not been any significant changes in their medical condition or medications for the preceding 6 weeks. Classification of renal impairment will be based using an MDRD equation
* Male subjects who are sexually active must use a condom and their partner if of childbearing potential must use a reliable method of contraception from the first dose of investigational product until 3 months after their last dose
* Have a body mass index (BMI) between 19 and 32 kg/m2 and weigh at least 50 kg

Exclusion Criteria:

* History of any clinically significant medical, neurologic or psychiatric disease or disorder (other than those previously defined as acceptable for this population, see inclusion criterion 1) which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results of the subject's ability to participate in the study: This includes seizure activity and repeated episodes of major depression
* Significant cardiovascular or cerebrovascular disease such as: a history of acute coronary syndrome; angina that has been symptomatic in the last 6 months; significant symptomatic arrhythmia; a stroke; transient ischemic attack that have occurred in the last 6 months
* History or presence of gastrointestinal or hepatic disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* Subjects who have type 2 diabetes must have an HbA1c of less than 8% according to the National Glycohemoglobin Standardization Program (NGSP) at screening
* Significant renal insufficiency as defined by eGFR per the MDRD formula <50 mL/min/1.73 m2 (individual eGFR measurements will be documented in the protocol).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse events | Range of 5 days
Neurological examinations | Range of 5 days
Visual acuity tests | Range of 5 days
Vital signs | Range of 5 days
Physical examinations | Range of 5 days
Laboratory parameters | Range of 5 days
Suicidality as assessed by the Columbia-Suicide Severity Rating Scale | Range of 5 days
Electrocardiograms | Range of 5 days

SECONDARY OUTCOMES:
Pharmacokinetic variables of TC-5214 by assessment of drug concentrations in plasma | Range of 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Hans A Eriksson, MD, Study Director — AstraZeneca; Wolfgang Kuhn, MD, Principal Investigator — Quintiles Phase 1; Aslak Rautio, MD, Principal Investigator — Quintiles Hermelinen
Locations (1):
- Research Site, Uppsala, Uppsala County, Sweden

REFERENCES:
- [Derived] Xu H, Henningsson A, Alverlind S, Tummala R, Toler S, Beaver JS, Al-Huniti N. Population pharmacokinetics of TC-5214, a nicotinic channel modulator, in phase I and II clinical studies. J Clin Pharmacol. 2014 Jun;54(6):707-18. doi: 10.1002/jcph.264. Epub 2014 Jan 16. PMID 24408516